CLINICAL TRIAL: NCT02659761
Title: A Prospective, Single Arm, Open-label 96 Week Observational Trial of the Tolerability, Adherence and Efficacy of a Dolutegravir/Abacavir/Lamivudine Single Tablet Regimen in HIV-1 Antibody Positive People Living With HIV With a History of Injection Drug Use Switching From Existing ART or Starting Treatment After Discontinuation of ART
Brief Title: Triumeq As an Integrase Single Tablet Regimen in People With HIV Who Inject Drugs
Acronym: TAISTR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision due to slow recruitment rates and no future recruitment foreseen
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAISTR_2016
Record Dates: First submitted 2016-01-08; First posted 2016-01-20 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; Injection drug use; Single-tablet antiretroviral treatment; Dolutegravir; Tolerability; Adherence; Efficacy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dolutegravir/abacavir/lamivudine (Experimental): All study subjects will receive triumeq (600 mg abacavir, 50 mg dolutegravir and 300 mg lamivudine) single tablet that will be taken orally, once daily, during 96 weeks
  Interventions: Drug: dolutegravir/abacavir/lamivudine

INTERVENTIONS:
Drug: dolutegravir/abacavir/lamivudine — 600 mg abacavir, 50 mg dolutegravir and 300 mg lamivudine single tablet taken orally, once daily, during 96 weeks
  Other Names: Triumeq

SUMMARY:
The purpose of this study is to assess the tolerability, adherence and efficacy of single tablet dolutegravir/abacavir/lamivudine antiretroviral therapy in people living with HIV with a history of injection drug use (IDU) switching from existing antiretroviral therapy (ART) or starting treatment after discontinuation of ART.

DETAILED DESCRIPTION:
Dolutegravir (DTG) is an integrase strand transfer inhibitor (INSTI) that supports once-daily dosing without the need for pharmacokinetic boosting and may be co-formulated with other antiretrovirals into a single-tablet regimen (STR). With people living with HIV with injection drug use (IDU) being more prone to unplanned antiretroviral therapy (ART) discontinuation and suboptimal adherence, DTG offers a high genetic barrier to resistance, a profile that reduces drug-drug interactions, with better tolerability and its availability as single tablet regimen (STR) combined with abacavir and lamivudine (ABC/3TC) is likely to improve adherence.

The aims of this study include:

* To assess tolerability through self-reported adverse effects and directed symptom questionnaire
* To determine change in number and severity of reported ART-related adverse effects from baseline to week 48 and 96
* To determine change in health-related quality of life (HRQOL) from baseline to week 48 and 96
* To determine change in frailty score from baseline to week 48 and 96
* To determine the percentage of subject with unscheduled ART discontinuations/ interruptions over 96 weeks
* To determine the estimated number of weeks of missed ART over 48 and 96 weeks of follow-up
* To determine change from baseline of medication possession ratio (MPR) at 48 and 96 weeks or adherence score as measured by an antiretroviral therapy medication self-report form at the same time points
* To determine the percentage of subjects with HIV RNA<40 copies/mL at 96 weeks
* To determine change in genotypic resistance profiles in subjects experiencing virological failure
* To determine change in CD4+ T-cell counts through 96 weeks
* To determine change in bone mineral density through 96 weeks
* To determine the number of subjects with any adverse and any serious adverse events (SAE) from baseline to week 96
* To determine the number of subject with Grade 1 to 4 laboratory abnormalities from baseline to week 96

This is a prospective, single arm, open-label 96 weeks clinical trial. Study subjects will be followed for 96 weeks post enrolment, with regular clinical evaluations, laboratory evaluations, safety and adherence assessment, quality of life and bone mineral density (BMD) measured at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults (≥18 years of age) with a history of IDU as the principal HIV transmission risk factor or with current or recent (past 12 months) history of IDU
* Either currently receiving an antiretroviral regimen but experiencing adherence or tolerability issues on current ART or restarting ART after an unscheduled treatment interruption
* Willing to switch current ART regimen
* No documented viral resistance to currently licensed HIV-1 integrase inhibitors, abacavir and lamivudine based either on previous HIV-1 genotypic resistance testing or in the judgment of the study investigators
* Integrase inhibitor naïve (defined as no-prior exposure to any INSTI)
* Documented negative HLAB*5701 allele

Exclusion Criteria:

* Subjects with active hepatitis B infection (defined as hepatitis B surface antigen (sAg) positive)
* Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification;
* Chronic renal failure estimated by glomerular filtration rate (eGFR) <60mls/min/1.73m2 at screening using the abbreviated Modification of Diet in Renal Disease (MDRD) equation
* Any active illness (including AIDS-defining illness) which in the opinion of the investigator would prevent the subject from completing all study assessments
* Female subjects who are pregnant, breastfeeding or planning future pregnancies or unwilling to take measures to avoid pregnancy for the study duration
* Any grade 4 laboratory abnormalities
* Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification
* Subjects weighing less than 40 kilograms and those are likely to require a Triumeq dose adjustment
* History or presence of allergy to the study drug or their components
* A diagnosis of cancer under current active chemotherapy or radiotherapy or having received chemotherapy or radiotherapy for a diagnosis of cancer within the previous 21 days prior to screening
* Subjects with a documented HLAB*5701 positive test on archived or screening bloods
* Concurrent use of any contraindicated medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Tolerability as assessed by the number of subjects with treatment-related adverse events measured using a self-reported form and directed symptoms questionnaire | Measured through 96 weeks
Proportion of subjects with unscheduled discontinuation of study treatment | Measured through 96 weeks
Change in medication possession ratio (MPR) at 48 weeks or adherence score as measured by an antiretroviral therapy medication self-report form | Measured through 48 weeks
Proportion of subjects with HIV RNA<40 cps/ml at 48 weeks | Measured through 48 weeks

SECONDARY OUTCOMES:
Change in number and severity of ART-related adverse effects | Measured through 48 weeks; 96 weeks
Change in health-related quality of life (HRQOL) | Measured through 48 weeks; 96 weeks
Change in frailty score | Measured through 48 weeks; 96 weeks
Estimated number of weeks of missed ART | Measured through 48 weeks; 96 weeks
Change from baseline in medication possession ratio (MPR) at 96 weeks or adherence score as measured by an antiretroviral therapy medication self-report form | Measured through 96 weeks
Proportion of subjects with HIV RNA<40 copies/mL | At 96 weeks
Change in the number of drug resistant mutations in subjects experiencing virological failure | Measured through 96 weeks
Change in bone mineral density | Measured through 96 weeks
Number of subjects with any adverse and any serious adverse events (SAE) and/or grade 1 to 4 laboratory abnormalities | Measured through 96 weeks
Change in CD4+ T-cell count | Measured through 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Mallon, MB BCh, PhD, FRCPI, Principal Investigator — University College Dublin
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

REFERENCES:
- [Background] Cohn SE, Jiang H, McCutchan JA, Koletar SL, Murphy RL, Robertson KR, de St Maurice AM, Currier JS, Williams PL. Association of ongoing drug and alcohol use with non-adherence to antiretroviral therapy and higher risk of AIDS and death: results from ACTG 362. AIDS Care. 2011 Jun;23(6):775-85. doi: 10.1080/09540121.2010.525617. PMID 21293986
- [Background] Meemken L, Hanhoff N, Tseng A, Christensen S, Gillessen A. Drug-Drug Interactions With Antiviral Agents in People Who Inject Drugs Requiring Substitution Therapy. Ann Pharmacother. 2015 Jul;49(7):796-807. doi: 10.1177/1060028015581848. Epub 2015 Apr 22. PMID 25902733
- See also: Centre for Experimental Host Pathogen Research — https://www.ucd.ie/medicine/research/researchcentres/ucdcentreforexperimentalpathogenhostresearch/